CLINICAL TRIAL: NCT01825993
Title: RANDOMISED STUDY ABOUT POTSOTERATORY PAIN CONTROL IN LAPAROSCOPIC SIGMOIDECTOMY
Brief Title: RANDOMISED STUDY OF EPIDURAL VS MPCA MORPHINE VS TAPP IN LAPAROSCOPIC SIGMOIDECTOMY
Acronym: 2013/004
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, LAURA MORA LOPEZ, General Surgeon, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIR TAP 2013; 2013-000556-17 (EudraCT Number)
Record Dates: First submitted 2013-03-29; First posted 2013-04-08 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Sigmoidal Tumour
Keywords: Peridural catheter; Morphine PCA; Transabdominal Block; laparoscopic sigmoidectomy
MeSH Terms: interventions — Levobupivacaine; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PCA endovenous (Experimental): 1mg/10 min Morphine
  Interventions: Drug: MORPHINE
- PERIDURAL CATHETER (Active Comparator): Peridural L-bupivacaine 0.25%
  Interventions: Drug: L-BUPIVACAINE ; MORPHINE
- TANSABDOMINAL BLOCK (TAP) (Active Comparator): L-BUPIVACAINE im
  Interventions: Drug: L-BUPIVACAINE ; MORPHINE

INTERVENTIONS:
Drug: L-BUPIVACAINE ; MORPHINE
  Other Names: PERIDURAL L-BUPIVACAINE; PCA MORPHINE
  Arms: PERIDURAL CATHETER; TANSABDOMINAL BLOCK (TAP)
Drug: MORPHINE
  Arms: PCA endovenous

SUMMARY:
The investigators would study the control of postoperative pain with peridural catheter, morphine PCA ev or Transabdominal block.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18
* Laparoscopic sigmoidectomy
* Informed consent firmed

Exclusion Criteria:

* ASA IV
* Urgent surgery
* Sigmoid tumour stage IV
* Cronic pain treatment
* No informed consent firmed
* Paliative surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
EVA (POSTOPERATIVE PAIN) | 72 H POSTOPERATIVE
  The investigators asked the patient the postoperative pain during teh first 72 hours by EVA scale.

SECONDARY OUTCOMES:
ADVERSE EFFECTS | five days
  the investigators look for adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: PUJOL GEMMA, MD, Principal Investigator — Corporacion Parc Tauli
Locations (2):
- Spain (2):
  - Corporacion Parc Tauli, Sabadell, Sabadell-Barcelona
  - Corporacion Parc Tauli, Sabadell, Sabadell-barcelona